CLINICAL TRIAL: NCT01773330
Title: High Resolution Manometry: Optimizing the Swallow Protocol
Brief Title: High Resolution Manometry for Swallowing
Acronym: HRM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study has been halted per PI and IRB recommendation
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 502-2012
Record Dates: First submitted 2013-01-11; First posted 2013-01-23 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Motility Disorder
Keywords: high resolution manometry; provocative swallow; impedence
MeSH Terms: interventions — gatorade; Supine Position; Sitting Position; Standing Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- esophageal manometry (Experimental): Esophageal manometry will be performed by swallowing different amounts of Gatorade depending on the protocol being followed. There will be alternate assignment of positions: supine position, semi-recumbent position,sitting position and standing up position.
  Interventions: Procedure: esophageal manometry; Dietary Supplement: Gatorade; Other: Supine position; Other: Semi-recumbent position; Procedure: Sitting; Procedure: Standing

INTERVENTIONS:
Procedure: esophageal manometry — Esophageal manometry will be performed by swallowing different amounts of Gatorade depending on the protocol being followed.There will be alternate assignment of positions: supine position, semi-recumbent position,sitting position and standing up position.
Dietary Supplement: Gatorade — The patient will be given Gatorade to drink at various times during the study.
Other: Supine position — Esophageal manometry will be performed by swallowing different amounts of Gatorade depending on the protocol being followed. There will be alternate assignment of positions: supine position, semi-recumbent position,sitting position and standing up position.
  Other Names: Semi-recumbent; Sitting; Standing up
Other: Semi-recumbent position — Esophageal manometry will be performed by swallowing different amounts of Gatorade depending on the protocol being followed. There will be alternate assignment of positions: supine position, semi-recumbent position,sitting position and standing up position.
  Other Names: Supine position; Sitting position; Standing up
Procedure: Sitting — Esophageal manometry will be performed by swallowing different amounts of Gatorade depending on the protocol being followed. There will be alternate assignment of positions: supine position, semi-recumbent position,sitting position and standing up position.
  Other Names: Supine; Semi-recumbent; Standing
Procedure: Standing — Esophageal manometry will be performed by swallowing different amounts of Gatorade depending on the protocol being followed. There will be alternate assignment of positions: supine position, semi-recumbent position,sitting position and standing up position.
  Other Names: Supine position; Semi-recumbent position; Sitting position

SUMMARY:
This study is using a new technology known as high resolution manometry which is used to evaluate patients that have trouble swallowing or have chest pain that is not related to the heart. The investigator wants to learn how the different positions of the body, in a lying position, semi-recumbent, sitting position or standing up, and the amount of liquid affects the outcome of the test. This will help the investigator to determine a standardized protocol for patients with trouble swallowing.

DETAILED DESCRIPTION:
The esophageal manometry will be performed in the motility lab at the Shands Endoscopy Center by passing a small tube into the patients nose, down the food pipe and into the stomach. The participants will be instructed to swallow a determined volume of Gatorade,depending on the protocol being followed. All participants will be starting in the supine position followed by semi-recumbent,sitting, then standing up. When the esophageal manometry is finished, the tube is removed and participation in this study is complete.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Healthy Volunteer
* No clinical evidence of dysphagia

Exclusion Criteria:

* History of prior dysphagia
* Prior esophageal or gastric dysmotility secondary to systemic conditions (scleroderma or diabetes mellitus)
* Known gastrointestinal malignancy
* Use of medications known to affect esophageal or gastric motility (e.g. anticholinergics, opiates, calcium channel blockers)
* Previous esophageal or gastric surgery
* Significant cardiac or respiratory disease
* Pregnancy (a pregnancy test will be performed in women of child-bearing potential)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Normal values for HRM while the patient is in the most physiologic position to stimulate normal eating habits. | up to 1 hour
  The patient is instructed to swallow a determined volume of Gatorade. All participants will be starting in the supine position followed by semi-recumbent,sitting, then standing up.

SECONDARY OUTCOMES:
Normal HRM values for a 200 ml provocative swallow. | up to 5 minutes
  The patient is instructed to swallow 200 ml of Gatorade in the sitting position.
Bolus clearance for each swallow with impedance. | up to 1 hour
  The patient is instructed to swallow a determined volume of Gatorade. All participants will be starting in the supine position followed by semi-recumbent,sitting, then standing up.
Normal size and diameter of esophagus and esophageal distension on a regular basis with the provocative swallow and impedance. | up to 1 hour
  The patient is instructed to swallow different amounts of Gatorade. All participants will be starting in the supine position followed by semi-recumbent,sitting, then standing up.
Standardization of the testing protocol for HRM and the reliability of volume and number of swallows. | up to 1 hour
  The patient is instructed to swallow different amounts of Gatorade. All participants will be starting in the supine position followed by semi-recumbent,sitting, then standing up.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhang, M.D., Ph.D., Principal Investigator — University of Florida
Locations (1):
- Shands Endoscopy Center, Gainesville, Florida, United States